CLINICAL TRIAL: NCT06379464
Title: Screening of New Markers of Gut Microbiota in Stroke and Depression: a Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CALM2303
Record Dates: First submitted 2024-04-06; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-08

CONDITIONS: Acute Ischaemic Stroke; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, urine, stool, mouth swab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with acute ischaemic stroke: Patients who met the diagnostic criteria of the 2018 Chinese guidelines for the diagnosis and treatment of acute ischemic stroke.
- Depressed patients: Patients who met the depression related criteria in the Chinese classification and diagnostic criteria for mental disorders.

SUMMARY:
Objectives of Study： Through the cross-sectional study of stroke and depression, key biomarkers are targeted by screening disease-associated intestinal bacteria, metabolites and immune factors through multi-omics techniques.

DETAILED DESCRIPTION:
With environmental changes, population aging, and the accelerated pace of social life, cerebrovascular diseases and mental illnesses have gradually become a major disease burden in China. Stroke is the second leading cause of death globally, as well as the leading cause of death and disability in China. In recent years, the prevalence and incidence of stroke have increased significantly in our country. Global Burden of Disease 2017 reported a stroke incidence rate of 258 (95% CI, 234-284) per 100,000 person-years and a mortality rate of 88 (95% CI, 80-94) per 100,000 person-years. Depression is one of the most common psychiatric disorders, with a lifetime prevalence of 15-18%, a recurrence rate of approximately 80%, and a disease outcome that worsens with increasing age of onset. World Health Organization measurements show that the disease burden of depression accounts for 10% of the total burden of all types of illness and disability. Its pathogenesis is still unknown, treatment options are limited, and most patients suffer from recurrent or prolonged illness for life. The etiology and pathophysiological mechanisms of stroke and depression remain unknown, and objective and reliable biological diagnostic markers are lacking.

As research strategies focusing on the central nervous system have encountered difficulties, the field has begun to look to the periphery for new clues. With the advancement of multi-omics studies integrating genome, transcriptome, epigenome, proteome, and metabolomics, important roles of gut microbiota have been discovered to influence the function and structure of the nervous system by regulating metabolites, the immune system, and neurotransmitters, etc. Benakis et al. found that gut-derived IL17+γδ T cells migrate to the meninges and promote post-stroke injury. Clearance of gut microbiota induced changes in dendritic cell activity, increased Treg cells, and decreased IL17+γδ T cells, which in turn alleviated stroke injury. Therefore, T-lymphocytes dependent on intestinal immunity are strongly associated with stroke severity. Previous studies have shown that IL-17 produced by γδ T cells in the meninges is an important factor in inducing anxious behavior and IFN-γ is important in maintaining social willingness, whereas pro-inflammatory factors such as IL-1β, IL-6 and TNF-α produced by inflammatory responses are highly correlated with depression, so that T-cell immunity may be associated with depression. Stroke and depression present a similar pathogenesis and spectrum of disease traits. IL-17+γδ T cells have been shown to be involved in the mechanism of injury after ischemic stroke; high levels of IL-17 are associated with depression, which is a common comorbidity of diseases such as the above. This suggests that the relevant immune pathways represented by IL-17 and γδ T cells may be a common pathogenic mechanism for stroke and depression. Previous studies have also shown that both diseases exhibit enrichment of Enterobacteriaceae. The applicant's team's findings, published in Gut, reveal that ischemic stroke can trigger a disturbance of the gut microbiota characterized by an overproliferation of Enterobacteriaceae, and that the disturbed microbiota can further contribute to the progression of brain injury and is associated with poor stroke outcomes. The mechanism is that stroke-induced intestinal ischemia leads to an increase in nitrate concentration in the intestinal mucus layer, and Enterobacteriaceae, which can undergo nitrate respiration, overpopulate as a result. A systematic review published in Clinical Psychology Review summarized 26 studies, including 20 case-control studies, and found that the gut microbiota of patients with anxiety and depression exhibited an enrichment of pro-inflammatory bacteria such as Enterobacteriaceae. Thus, disorders of the gut microbiota characterized by Enterobacteriaceae are all associated with the above major brain diseases.

In summary, stroke and depression patients share common and respective unique characteristics of gut microbiota, metabolites, and immune factors. In this study, we intend to identify the key factors of intestinal bacteria and target novel biomarkers in stroke and depression through cross-sectional study of stroke and depression, using cutting-edge multi-omics technology.

ELIGIBILITY:
AIS Patients:

Inclusion Criteria:

1. Age range from 18 to 90 years old;
2. Patients who met the diagnostic criteria of the 2018 Chinese guidelines for the diagnosis and treatment of acute ischemic stroke;
3. Sign the informed consent form, provide relevant medical history information and provide blood, urine and stool samples.

Exclusion Criteria:

1. Serious systemic diseases including malignancies;
2. Alanine aminotransferase or aspartate aminotransferase >2 times the upper limit of normal value or severe liver disease;
3. Creatinine >1.5 times the upper limit of normal or severe nephropathy;
4. A long-term history of drinking, drug taking and chemical poisoning. A long-term history of drinking refers to a history of more than 5 years, equivalent to alcohol >40g/d for men and 20g/d for women, or a history of heavy drinking within 2 weeks, equivalent to alcohol >80g/d;
5. Those with previous history of intestinal tumor, irritable bowel syndrome or inflammatory bowel disease or diagnosed in Hospital;
6. Unable to retain the required samples.

Depressed patients:

Inclusion Criteria:

1. Age range from 18 to 90 years old;
2. Patients who met the depression related criteria in the Chinese classification and diagnostic criteria for mental disorders;
3. Sign the informed consent form, provide relevant medical history information and provide oral swabs, blood, urine and stool samples.

Exclusion Criteria:

1. Serious systemic diseases including malignancies;
2. Alanine aminotransferase or aspartate aminotransferase >2 times the upper limit of normal value or severe liver disease;
3. Creatinine >1.5 times the upper limit of normal or severe nephropathy;
4. A long-term history of drinking, drug taking and chemical poisoning. A long-term history of drinking refers to a history of more than 5 years, equivalent to alcohol >40g/d for men and 20g/d for women, or a history of heavy drinking within 2 weeks, equivalent to alcohol >80g/d;
5. Those with previous history of intestinal tumor, irritable bowel syndrome or inflammatory bowel disease or diagnosed in Hospital;
6. Unable to retain the required samples.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients with acute ischaemic stroke；
  2. Depressed patients
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The severity of neurological damage in stroke patients | The evaluation will be conducted on the second day after admission
  The severity of neurological damage in stroke patient evaluated by National Institutes of Health Stroke Scale(NHISS), the scoring range is 0-42 points, with higher scores indicating more severe neurological damage.
The functional recovery outcomes after stroke | The evaluation will be conducted at 3 months after admission
  The functional recovery outcomes after stroke evaluated by Modified Rankin Scale(mRS), the scoring range is 0-6 points, with higher scores indicating worse functional outcome.
The severity of symptoms in patients with depression | The evaluation will be conducted on the second day after admission
  The severity of symptoms in patients with depression is evaluated by Hamilton Depression Scale(HAMD), the scoring range is 0-54 points, with higher scores indicating more severe depressive states.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, Study Chair — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guanzhou, Guangdong, China